CLINICAL TRIAL: NCT01351766
Title: Behavioral Activation Intervention, Reward Processing, and Youth Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Laura MacPherson, Study Principal Investigator, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA029445; R21DA029445 (NIH)
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Smoking
Keywords: Behavioral Activation
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Activation for Smoking (Experimental): Eight 60-minute group sessions over an eight-week period. Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue after treatment sessions have ended.
  Transdermal Nicotine: Participants will use 8 weeks of the nicotine patch at 24 hour doses of 21, 14, and 7 mg respectively depending on participant's initial level of nicotine use. Nicotine patch dose will decrease at 2 or 4 week increments also specific to participant's initial nicotine level.
  Interventions: Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Drug: Transdermal Nicotine Patch — Transdermal Nicotine: Participants will use 8 weeks of the nicotine patch at 24 hour doses of 21, 14, and 7 mg respectively depending on participant's initial level of nicotine use. Nicotine patch dose will decrease at 2 or 4 week increments also specific to participant's initial nicotine level.
  Other Names: Nicoderm CQ

SUMMARY:
The primary purpose of this study is to develop a specialized behavioral activation treatment for smoking in youths ages 18-21 with elevated depressive symptoms. In the first phase we utilize focus groups and pilot testing with 15 youths to develop the behavioral activation smoking treatment for youth. In Phase II, we will conduct an open-label trial of the new treatment that will include 8 weeks of transdermal nicotine patch, which will begin at the time of quitting smoking. Participants will be followed over 26 weeks post-quit date. A subset of participants will also undergo an fMRI session to examine reward sensitivity.

DETAILED DESCRIPTION:
1. 18-21 years of age,
2. a regular smoker for at least 6 months
3. currently smoking an average of at least 5 cigarettes per day
4. want to quit smoking
5. report current elevated depressive symptoms

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 21 years of age
* a regular smoker for at least 6 months
* currently smoking an average of at least 5 cigarettes per day
* want to quit smoking
* report current elevated depressive symptoms

Exclusion Criteria:

* current Axis I disorder
* psychoactive substance dependence (excluding nicotine dependence) within the past 6 months
* current use of psychotropic medication or participation in any form of psychotherapy
* a history of significant medical condition (e.g., cardiovascular , neurological, gastrointestinal), pregnancy and/or breast feeding, or other systemic illness
* limited mental competency [Mini Mental State Examination score < 23] and/or the inability to give informed, voluntary, written consent to participate
* current use of any pharmacotherapy for smoking cessation not provided by the researchers during the quit attempt

Additional Exclusion criteria only for the fMRI portion:

* cerebrovascular disease
* high blood pressure
* diabetes
* use of psychotropic medications in 3 weeks prior to participation in fMRI protocol
* exposure to extreme trauma
* lifetime history of mania, psychosis, or pervasive developmental disorder,
* being ambidextrous or left handed
* any metal implants, heart pacemaker, permanent retainer
* tattoos containing metal dyes
* claustrophobia.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura MacPherson, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, College Park, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Activation for Smoking: * Eight, 60-minute group sessions over an 8 week period
  * Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking, and will continue after treatment sessions have ended
Period: Overall Study
Arm/Group | Behavioral Activation for Smoking
Started | 39
Completed | 36
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Analysis population is not different from the assignment in Participant Flow.
Groups:
- Behavioral Activation for Smoking: Behavioral Activation for Smoking (BATSY) includes standard smoking cessation strategies and identifying life areas, values, and daily activities to help manage mood. Participants will complete between group exercises and will also monitor and plan daily activities in line with their values. Treatment will be delivered in 8, 60-minute group sessions over an 8-week period. Participants will also be provided 8 weeks of the transdermal nicotine patch.
  Transdermal Nicotine Patch: 8 weeks of the Transdermal Nicotine Patch Nicoderm CQ at 24 hour doses of 21, 14, and 7 mg respectively depending on participant's initial level of nicotine use. Nicotine patch dose will decrease at 2 or 4 week increments also specific to participant's initial nicotine level.
Arm/Group | Behavioral Activation for Smoking
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.00 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Smoking-Abstinent for 7 Days, 12 Weeks Post Quit Date
Description: 7 days of smoking abstinence confirmed via expired carbon monoxide at 12 weeks
Time Frame: 12 weeks post quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation for Smoking
Number analyzed (Participants) | 39
Participants | 7

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 20 weeks.
Description: Definition of adverse event and/or serious adverse event does not differ from clinicaltrials.gov definitions.
Arm/Group | Behavioral Activation for Smoking
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No